CLINICAL TRIAL: NCT04285840
Title: Arterial Versus Venous Activated Clotting Time Measurements During Atrial Fibrillation Ablations
Brief Title: Arterial Versus Venous Activated Clotting Time (ACT) Measurements During Atrial Fibrillation Ablations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00104539
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): To establish a standardized procedure for venous ACT sampling during atrial fibrillation ablation. Analyses will examine the relationship and agreement between venous and arterial ACTs.
  Interventions: Other: Venous ACT

INTERVENTIONS:
Other: Venous ACT — Matched/paired venous ACT samples will be drawn at the same time as arterial ACT samples to compare the results agreement between venous and arterial ACTs. Subjects undergoing atrial fibrillation ablations will continue to have Heparin dosed on the arterial ACT sample results only per the standard of care. Heparin will not be administered based on venous ACT levels obtained during this study.

SUMMARY:
Activated clotting times (ACTs) are routinely measured throughout atrial fibrillation ablations to monitor anticoagulation prior to and after heparin administration. Routinely, ACTs are obtained from an arterial line established prior to heparin administration. With technological advances, the cardiac intervention team is interested in eliminating the need for arterial lines for noninvasive monitoring devices; eliminating arterial lines could decrease the risk of bleeding, infection, and pain. Since procedural access requires femoral vein catheterization, obtaining ACTs through the venous sheath would not pose additional risks to the patient. In this study it proposed to draw paired arterial and venous ACT samples in ablation procedures to compare the agreement between venous and arterial ACTs for adequate patient treatment planning.

DETAILED DESCRIPTION:
This project aims to establish a standardized procedure for venous ACT sampling during atrial fibrillation ablation in 50 adults. Analyses will examine the relationship and agreement between venous and arterial ACTs. It is anticipated that the standardized procedure could eliminate the need for an arterial line for ACT measurement which would reduce patient risks for bleeding, infection, and discomfort.

Patients who are scheduled for for atrial fibrillation ablations will be invited to participate in this project. An information sheet will be provided about the project to potential participants. If the potential participant expresses interest, a study specific consent consent will be obtained to allow the additional paired blood samples to be drawn throughout the procedure. The additional blood volume to be drawn is expected to be less than or equal to a teaspoon of venous blood. Participation will be completely voluntary.

Patients will undergo usual standard of care for the procedure, including usual arterial and venous sheath/catheter insertions. After obtaining venous and arterial access, baseline ACTs will be drawn using the outlined ACT sampling procedure. The ACT value for both arterial and venous samples will be obtained using the standard procedure for Hemochron Signature Elite point-of-care testing; this test uses less than 0.5 cc blood. ACT samples will be performed at baseline (pre-heparin administration), every 30 minutes during the procedure (per standard ACT monitoring protocol to obtain and maintain desired ACT), and at the end of procedure prior to arterial and venous sheath removal. Time of procedure ranges from 2 to 4 hours and may result in a minimum of 2 paired samples (pre and end) to a maximum of 9 paired samples (pre, end, and every 30 minutes) per patient; this equates to an additional 1 cc to 4.5 cc of additional blood for paired sampling per patient.

ACT arterial and venous sampling procedure: Using a stopcock at the nearest point of insertion, withdraw 30 cc of blood in a syringe; turn the stopcock and remove 0.5cc of blood for ACT testing; turn the stopcock to return the 30 cc blood and flush the line; remove the syringe with the ACT sample and flush the line with saline, replace syringes for the next ACT sampling process.

Patients undergoing atrial fibrillation ablations will continue to have Heparin dosed on the arterial ACT sample results only per the standard of care. Heparin will not be administered based on venous ACT levels obtained during this project. The purpose for paired sampling is to verify that the proposed venous sampling method is accurate and provides an evaluable sample to compare with the ACT sample results.

ELIGIBILITY:
Inclusion Criteria:

Adult scheduled for routine atrial ablation procedure

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of venous ACT samples that match arterial ACT sample results during atrial fibrillation ablation | Day of atrial fibrillation ablation procedure
  Paired samples pre and during the ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Allen Deborah, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke Health Raleigh, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No